CLINICAL TRIAL: NCT00314288
Title: A Multicenter, Multinational, Randomised, Double-blind, Placebo-controlled, Parallel-group, Dose-finding Study to Investigate the Anti-dyskinetic Efficacy and Safety of Sarizotan in Parkinson Patients With L-dopa-induced Dyskinesia
Brief Title: Sarizotan in Parkinson Patients With L-dopa-induced Dyskinesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMR 62225-006
Record Dates: First submitted 2006-04-12; First posted 2006-04-13 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Parkinson's Disease; Dyskinesia
Keywords: Parkinson's Disease; Dyskinesia; L-dopa-induced dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesias

INTERVENTIONS:
Drug: Sarizotan HCl

SUMMARY:
The primary purpose of the study is to investigate the anti-dyskinetic effect of several doses of sarizotan in Parkinson patients in order to generate information on the dose-response relationship (dose-finding).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* The subject is an out-patient
* Age 30 years or above
* Dyskinesias present during more than 25% of the waking day
* Dyskinesias at least moderately disabling
* Written informed consent

Exclusion Criteria:

* Pregnancy and/or lactation
* Participation in another study within the last 30 days
* Dementia or other psychiatric illness that prevents provision of informed consent
* History of allergic disorders such as asthma
* Known hypersensitivity to the study treatment(s)
* Known hypersensitivity to ACTH

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2002-07; Study Completion 2003-07

CONTACTS AND LOCATIONS:
Locations (51):
- United States (17):
  - Fountain Valley, California
  - Sunnyvale, California
  - Miami, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Augusta, Maine
  - Boston, Massachusetts
  - Kansas City, Missouri
  - Brooklyn, New York
  - New York, New York
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Pawtucket, Rhode Island
  - Memphis, Tennessee
  - Houston, Texas
- Leuven, Belgium
- Sofia, Bulgaria
- Canada (3):
  - Edmonton
  - Saskatoon
  - Vancouver
- France (5):
  - Clermont-Ferrand
  - Marseille
  - Nantes
  - Paris
  - Toulouse
- Germany (7):
  - Bochum
  - Dresden
  - Leipzig
  - Lübeck
  - München
  - Ulm
  - Wiesbaden
- Hungary (3):
  - Budapest
  - Győr
  - Miskolc
- Portugal (2):
  - Coimbra
  - Lisbon
- Romania (3):
  - Bucaresti
  - Constanța
  - Târgu Mureş
- South Africa (5):
  - George
  - Plumstead Cape Town
  - Rosebank
  - Sunninghill
  - Wilgers
- United Kingdom (4):
  - Cambridge
  - Newcastle
  - Nottingham
  - Sheffield